CLINICAL TRIAL: NCT03531424
Title: On-Site Augmented-Reality Computed Tomography Plus Angiography Versus Angiography Alone for Guiding Percutaneous Coronary Intervention in Native Coronary Lesions - Randomized Study
Brief Title: Augmented-Reality CTA Plus Angiography vs Angiography Alone for Guiding PCI in Coronary Lesions - Randomized Study
Acronym: AR-PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul Knaapen (Other)
Responsible Party: Sponsor-Investigator, Paul Knaapen, Clinical Professor, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL63928.029.17
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Stenosis; Percutaneous Coronary Intervention; Stents; Computed Tomography Angiography; Augmented Reality
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiographic guided PCI (Active Comparator): Angiographic guided PCI is coronary revascularization based on stand-alone angiography.
  Interventions: Procedure: Angiographic guided PCI
- CTA guided PCI (Experimental): CTA guided PCI is coronary revascularization based on systematic use of CTA plus coronary angiography.
  Interventions: Procedure: Augmented-Reality CTA guided PCI

INTERVENTIONS:
Procedure: Angiographic guided PCI — Angiographic guided PCI is coronary revascularization based on stand-alone angiography.
  Arms: Angiographic guided PCI
Procedure: Augmented-Reality CTA guided PCI — Augmented-Reality CTA guided PCI is coronary revascularization based on systematic use of CTA datasets displayed in augmented-reality glass plus coronary angiography.
  Arms: CTA guided PCI

SUMMARY:
The purpose of this study is to compare revascularization strategy and its immediate results after augmented-reality computed tomography angiography (CTA) guided vs. standard angiography guided percutaneous coronary intervention (PCI) in native coronary lesions.

DETAILED DESCRIPTION:
While stand-alone angiography is the first-line imaging modality for guidance of PCI, it has some inherent limitations which may result in suboptimal stent placement related to residual reference segment disease and stent underexpansion. Coronary CTA, on the other hand, can provide reliable measurements of the vessel size and lesion length as well as the visualization of the morphological features of coronary plaque, and has been suggested as potentially valuable for changing PCI technique. The AR-PCI trial has been designed as a single-center, investigator initiated and investigator sponsored, randomized (1:1), controlled, prospective clinical trial. It is hypothesized that the review of CTA datasets using augmented-reality glass in the catheterization laboratory could influence PCI treatment strategy and its immediate results by more adequate lesion coverage with less residual disease and better stent expansion as compared to traditional angiography-guided PCI alone.

ELIGIBILITY:
Inclusion Criteria:

* patients with documented obstructive CAD defined as the presence of at least 1 stenosis ≥70% in a native coronary artery in whom PCI is considered based on clinical grounds

Exclusion Criteria:

* refusal or inability to provide written informed consent
* subjects in whom the quality of coronary CTA is insufficient
* bifurcation lesions, by which strategies other than a single cross-over stent technique are anticipated
* left main coronary artery stenosis
* chronic total occlusion
* in-stent restenosis
* chronic renal failure (estimated glomerular filtration rate <30 ml/min)
* known allergy to contrast
* untreated hyperthyroidism
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Stent length | 1 day
  Length of the stented segment
Predicted stent diameter | 1 day
  Predicted final stent diameter according to a compliance chart

SECONDARY OUTCOMES:
Nominal stent diameter | 1 day
  Nominal diameter of the implanted stent
Number of stents | 1 day
  Total number of stents
Predilation | 1 day
  Balloon predilation for lesion modification
Postdilation | 1 day
  Balloon postdilation for stent expansion
Maximal balloon pressure | 1 day
  Maximal balloon pressure applied during PCI
Maximal balloon diameter | 1 day
  Maximal balloon diameter applied during PCI
Stent-edge dissection | 1 day
  Stent-edge dissection by coronary angiography
Post-procedural residual diameter stenosis | 1 day
  Post-procedural residual diameter stenosis by 3D QCA
Post-procedural residual area stenosis | 1 day
  Post-procedural residual area stenosis by 3D QCA
Post-procedural minimum lumen diameter | 1 day
  Post-procedural minimum lumen diameter by 3D QCA
Post-procedural minimum lumen area | 1 day
  Post-procedural minimum lumen area by 3D QCA
Post-procedural lumen diameters at the reference segments | 1 day
  Post-procedural lumen diameters at the reference segments by 3D QCA
Post-procedural lumen areas at the reference segments | 1 day
  Post-procedural lumen areas at the reference segments by 3D QCA
Post-procedural volume of the stented segment | 1 day
  Post-procedural volume of the stented segment by 3D QCA
Post-procedural volume of the reference segments | 1 day
  Post-procedural volume of the reference segments by 3D QCA

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center Amsterdam, Amsterdam, De Boelelaan 1117, Netherlands

IPD SHARING:
Plan to Share IPD: No